CLINICAL TRIAL: NCT05665972
Title: Effects of Mandala Coloring on Premenstrual Syndrome: Randomized Controlled Experimental Study
Brief Title: Effects of Mandala Coloring on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Efsun Derin, Research Assistant, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliED-2
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; Mandala coloring
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala coloring group (Experimental): Mandala painting will be applied to women suffering from premenstrual syndrome.
  Interventions: Other: Mandala coloring
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce premenstrual syndrome symptoms.

INTERVENTIONS:
Other: Mandala coloring — Each participant will be given 12 colored felt-tip pen paint sets and 12 mandala coloring pages by the researchers. Participants will be asked to dye for 3 menstrual cycles, 14 days before the start of menstruation, 1 day a week, at any time of the day and for an average of 20-30 minutes each time.
  Arms: Mandala coloring group

SUMMARY:
This research was planned as a randomized controlled experimental study in order to reduce premenstrual syndrome symptoms of women with premenstrual syndrome.

DETAILED DESCRIPTION:
Occurs in the luteal phase and decreases or declines significantly with the onset of menstruation; physical such as breast tenderness, headache, bloating; Premenstrual syndrome is a health problem with more than 150 psychological and behavioral symptoms such as anger outbursts, irritability, anxiety, mood fluctuations, sleep and eating disorders.

Symptoms experienced during the premenstrual period lead to results such as mood/affective disorder in women, deterioration in daily life activities and social relations, an increase in negative health behaviors, as well as low academic performance in students, decreased participation in classes, getting low grades in exams, and not showing up for exams.Since its etiology is unclear, no specific treatment method can be found, and non-pharmacological therapies such as stress control, lifestyle changes, exercise and complementary therapies such as evening primrose oil, chasteberry and acupuncture are applied in its management.

Psychiatrist Carl Gustav Jung discovered the psychic healing transformations created by mandala painting, one of the art therapy methods, through his own experience and that of his patients.

Various studies have determined that mandala coloring improves physical and psychological symptoms, but no studies have been conducted with PMS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Fully answering survey and scale forms.
* Ability to read and understand Turkish
* Being between the ages of 18 and 30 years
* Having regular menstruation (between 21 and 35 days)
* Having 45 or more from PMSS

Exclusion Criteria:

* Unwilling to continue working
* Having any problem that prevents communication (such as hearing, speaking, and understanding abilities),
* Having a gynecological disease (abnormal uterine bleeding, uterine fibroids, ovarian cysts, hormonal treatment, etc.)
* Having a chronic or physical illness
* Having a mental illness
* Being under psychiatric treatment (Pharmacotherapy or psychotherapy)
* Taking medication for menopausal symptoms
* Using one of the pharmacological or non-pharmacological methods to reduce premenstrual symptoms (COCs, acupressure, homeopathy, etc.)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | between one to six months
  The form consists of questions about socio-demographic and menstrual periods.

SECONDARY OUTCOMES:
Premenstrual Syndrome Scale | between one to six months
  The Premenstrual Syndrome Scale was developed by Gençdoğan (2006) to measure premenstrual symptoms and determine their severity. It is a five-point Likert type scale (Never, Rarely, Sometimes, Frequently, Always) consisting of 44 items. The scale is scored as "Never" 1 point, "Rarely" 2 points, "Sometimes" 3 points, "Frequently" 4 points, and "Always" 5 points. The Premenstrual Syndrome Scale includes nine subdimensions which are depressive affect, anxiety, fatigue, irritability, depressive thoughts, pain, appetite change, sleep change, and bulge. The total Premenstrual Syndrome Scale score is obtained from the total points received from all nine subdimensions of the scale. A higher score from the scale means the intensity of Premenstrual Syndrome Scale symptoms increases too. The Cronbach's alpha coefficient of the scale was 0.75.

CONTACTS AND LOCATIONS:
Overall Officials: Efsun DERİN, Principal Investigator — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derin E, Solt Kirca A. The Effect of Mandala Coloring on Premenstrual Syndrome: A Randomized Controlled Experimental Study. Holist Nurs Pract. 2025 Nov 3. doi: 10.1097/HNP.0000000000000724. Online ahead of print. PMID 41177972